CLINICAL TRIAL: NCT05538026
Title: Efficacy and Safety of Fecal Microbiota Transplantation as add-on Therapy in Patients With Mild-To-Moderate Ulcerative Colitis: A Randomized, Clinical Trial
Brief Title: Effectiveness of Fecal Microbiota Transplantation as add-on Therapy in Mild-to-moderate Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Collaborators: Ukrainian Research and Practical Centre of Endocrine Surgery, Transplantation of Endocrine Organs and Tissues of the Ministry of Health of Ukraine (Unknown)
Responsible Party: Principal Investigator, Nazarii Kobyliak, Associate Professor, Endocrinology Department, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-UC
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Ulcerative Colitis Chronic Mild; Inflammatory Bowel Diseases
Keywords: Ulcerative Colitis; fecal microbiota transplantation; gut microbiota; dysbiosis; inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Dysbiosis | interventions — Mesalamine; Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care group (Active Comparator): mesalazine (Pentasa) at a daily dose of 3 g (2 g orally + 1 g rectally)
  Interventions: Drug: Mesalazine
- Fecal transplantation (Experimental): Fecal transplantation of fresh prepared feces from healthy donor. Application by colonoscope in proximal half of colon.
  Interventions: Biological: Fecal transplantation

INTERVENTIONS:
Drug: Mesalazine — daily dose of 3 g (2 g orally + 1 g rectally)
  Other Names: Pentasa
  Arms: standard care group
Biological: Fecal transplantation — Preparation of fresh feces by blending in 0.9 % saline and crude filtering. The solution is applied in proximal colon of UC patient by colonoscopy after standard bowel preparation.
  Arms: Fecal transplantation

SUMMARY:
Ulcerative colitis (UC) is a chronic immune-mediated inflammatory bowel disease (IBD) that almost always affects the rectum and often extends to the more proximal colon. UC usually begins at a young age (15-30 years), most patients (~ 85%) have a mild or moderate activity, characterized by periods of exacerbation and remission. Considering the important pathogenetic role of gut dysbiosis, recently, as an additional method of treating UC, it is considered a modification of altered gut microbiota using various drug and non-drug methods. One such method is fecal microbiota transplantation (FMT), consisting of the simultaneous replacement of the gut microbiota of a sick recipient with fecal material from a healthy donor. Even though so far the only officially approved indication for FMT is recurrent Clostridium difficile infection, however, the effectiveness of FMT is currently being studied in the treatment of other gastrointestinal and non-gastrointestinal pathologies, including UC. To date, several controlled and uncontrolled studies have been conducted to study the effectiveness of FMT in UC, showing encouraging results. This study aimed to assess the clinical and microbiological efficacy, tolerability, and safety of FMT as add-on therapy to basic therapy, in patients with mild-to-moderate UC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60;
* Endoscopically and morphologically confirmed UC;
* Negative results of stool culture for the presence of pathogenic bacteria (Shigella spp., Salmonella spp., Campylobacter spp., Yersinia spp.) and toxin-producing Clostridioides difficile;
* partial Mayo score of 4-6;
* Mayo endoscopic subscore ≥1;
* Fecal calprotectin > 150 mcg/g
* Treatment with mesalazine at a daily dose of 3 g during the last 4 weeks

Exclusion Criteria:

* Pregnancy, planning pregnancy or breastfeeding;
* Postponed operations on the abdominal cavity;
* Severe mental disorders, alcohol or drug abuse;
* Use of systemic corticosteroids, biological agents, and probiotics within 8 weeks before study
* Any condition or circumstance that would, in the opinion of the investigator, prevent completion of the study or interfere with analysis of study results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Change in partial Mayo score > 2 points | 8 weeks
  Partial Mayo score composed of four parts: rectal bleeding, stool frequency, physician assessment, and endoscopy appearance. Each part is rated from 0 to 3, giving a total score of 0 to 12. Partial Mayo score (eliminates endoscopy) and of 2 to 4 points indicates mildly active disease, a score of 5 to 6 points indicates moderately active disease, and a score of 7 to 9 points indicates severely active disease
Changes in fecal calprotectin | 8 weeks
  expressed in µg/g

SECONDARY OUTCOMES:
Microbiome profile change | 4 weeks
  Characterization of fecal microbiome by metagenomic analysis before and after intervention Characterization of fecal microbiome by metagenomic analysis before and after intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Ukraine (2):
  - Bogomolets National Medical University, Kyiv
  - Ukrainian Research and Practical Centre of Endocrine Surgery, Transplantation of Endocrine Organs and Tissues of the Ministry of Health of Ukraine, Kyiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tkach S, Dorofeyev A, Kuzenko I, Falalyeyeva T, Tsyryuk O, Kovalchuk O, Kobyliak N, Abenavoli L, Boccuto L. Efficacy and safety of fecal microbiota transplantation via colonoscopy as add-on therapy in patients with mild-to-moderate ulcerative colitis: A randomized clinical trial. Front Med (Lausanne). 2023 Jan 12;9:1049849. doi: 10.3389/fmed.2022.1049849. eCollection 2022. PMID 36714101